CLINICAL TRIAL: NCT03407222
Title: Effect of Monitoring and Education of Step Number Assessed by Smartphone Application on Blood Glucose, Weight and Blood Pressure in Patients With Type 2 Diabetes
Brief Title: Effect of Monitoring of Step Number on Diabetes
Acronym: PHR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jae Hyeon Kim, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-12-052
Record Dates: First submitted 2018-01-16; First posted 2018-01-23 (Actual); Last update posted 2019-03-25 (Actual); Status verified 2019-03

CONDITIONS: Type 2 Diabetes Mellitus; Physical Activity
Keywords: Type 2 Diabetes Mellitus; Physical Activity; Personal health record; Intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Intervention Model Description: Send text messages which encourage step-by-step increment of daily step count
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Intervention group receives weekly text messages which encourage the increment of daily step count
  Interventions: Other: Text messages
- Control group (No Intervention): Control group does not receive text message

INTERVENTIONS:
Other: Text messages — Text messages which encourage the increment of daily step count
  Arms: Intervention group

SUMMARY:
In this study, investigators measured the number of steps, blood pressure, blood glucose, and weight in daily life through the smartphone personal health record application for patients with type 2 diabetes. The efficacy of text message intervention, which encourages an increase in the number of steps per week for 12 weeks, on an increase in the number of daily steps and changes in glucose levels, weight, and blood pressure will be investigated. Also, the durability of intervention will be checked after 12 weeks of intervention ending.

DETAILED DESCRIPTION:
This clinical study is a single institution, randomized, prospective study and monitors the average daily number of steps per week using a smartphone personal health record application developed by Samsung Medical Center for patients with type 2 diabetes. The study subjects were divided into five groups such as 1) basal activity (<2500 steps/day), 2) limited activity (2500-4999 steps/day), 3) low activity (5000-7499 steps/day), 4) somewhat active (7500-9999 steps/day), 5) active (10000-12499 steps/day), 6) highly active (≥12500 steps/day)according to the average number of steps per day. During the 12-week period, the intervention group receives the text messages that encourage step-by-step increments every week, and the control group does not receive text messages. The effect of 12-week step monitoring and education on the change in daily step count will be analyzed. Also, the effect of change in daily step count on glucose level, body weight, and blood pressure will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 2 diabetes aged 20-69 years
* Patients with a HbA1c of less than 8.5% measured during screening (may be replaced by a test value within 3 months of screening visit )
* Patients who have not been prescribed diabetic medication for the past 4 weeks or who have taken more than one oral hypoglycemic agent for more than 12 weeks at a certain dose
* BMI ≥ 23 kg/m2
* Available for use Samsung Galaxy S4 or later Android smartphone and wireless internet
* Patients who voluntarily agreed to participate in this clinical study

Exclusion Criteria:

* Diabetes other than type 2 diabetes, including type 1 diabetes, gestational diabetes
* Patients who are taking insulin or GLP-1 agonist other than oral hypoglycemic agent
* Patients with uncontrolled chronic liver disease
* Patients with acute kidney injury
* Patients with psychological disorder
* Patients who are taking weight lowering agent
* Patients with alcohol or drug addiction within the last 3
* Patients who are taking systemic steroid
* Patients who are breastfeeding or pregnant
* Patients who did not voluntarily agree to the study
* Patients who are unsuitable for participation in clinical research

Ages: 20 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
change in daily step count after 12 weeks of intervention | Week 12
  change in daily step count after 12 weeks of intervention

SECONDARY OUTCOMES:
mean daily step count after 12 weeks of intervention | Week 12
  mean daily step count after 12 weeks of intervention
the proportion of patients who reach participant-day during the 12 weeks of intervention | Week 12
  the proportion of patients who reach participant-day during the 12 weeks of intervention The participant-day means the day the participant reach thier upper group of daily step count
mean daily step count at Week 24 | Week 24
  mean daily step count at Week 24
the proportion of patients who reach participant-day during the Week 13-24 | Week 24
  the proportion of patients who reach participant-day during the Week 13-24
the proportion of patients whose HbA1c levels <6.5% without severe hypoglycemia | Week 12
  the proportion of patients whose HbA1c levels <6.5% without severe hypoglycemia
the proportion of patients whose HbA1c levels <6.5% without severe hypoglycemia | Week 24
  the proportion of patients whose HbA1c levels <6.5% without severe hypoglycemia
HbA1c levels | Week 12
  HbA1c levels (%)
HbA1c levels | Week 24
  HbA1c levels (%)
Fasting glucose levels | Week 12
  Fasting glucose levels (mg/dL)
Fasting glucose levels | Week 24
  Fasting glucose levels (mg/dL)
Body weight | Week 12
  Body weight (kg)
Body weight | Week 24
  Body weight (kg)
Blood pressure | Week 12
  Blood pressure (mmHg)
Blood pressure | Week 24
  Blood pressure (mmHg)
IPAQ (international physical activity questionnaire) score | Week 12
  IPAQ (international physical activity questionnaire) score are consisted of 7 questions regarding frequency of exercise, intensity of exercise, and duration of exercise. Using its automatic report, the results can be calculated as weekly physical activity level (low, intermediate, high).
IPAQ (international physical activity questionnaire) score | Week 24
  IPAQ (international physical activity questionnaire) score are consisted of 7 questions regarding frequency of exercise, intensity of exercise, and duration of exercise. Using its automatic report, the results can be calculated as weekly physical activity level (low, intermediate, high).
number of recordings on personal health record application | Week 12
  number of recordings on personal health record application
number of recordings on personal health record application | Week 24
  number of recordings on personal health record application
Total cholesterol | Week 12
  Total cholesterol (mg/dL)
Total cholesterol | Week 24
  Total cholesterol (mg/dL)
High-density lipoprotein cholesterol | Week 12
  High-density lipoprotein cholesterol (mg/dL)
High-density lipoprotein cholesterol | Week 24
  High-density lipoprotein cholesterol (mg/dL)
Triglycerides | Week 12
  Triglycerides (mg/dL)
Triglycerides | Week 24
  Triglycerides (mg/dL)
low-density lipoprotein cholesterol | Week 12
  low-density lipoprotein cholesterol (mg/dL)
low-density lipoprotein cholesterol | Week 24
  low-density lipoprotein cholesterol (mg/dL)

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim G, Kim S, Lee YB, Jin SM, Hur KY, Kim JH. A randomized controlled trial of an app-based intervention on physical activity and glycemic control in people with type 2 diabetes. BMC Med. 2024 May 1;22(1):185. doi: 10.1186/s12916-024-03408-w. PMID 38693528